CLINICAL TRIAL: NCT00082576
Title: A Phase II/III, Randomized, Double-Blind, Comparative Trial Of Azithromycin Plus Chloroquine Versus Mefloquine For The Treatment Of Uncomplicated Plasmodium Falciparum Malaria In Africa
Brief Title: Azithromycin Plus Chloroquine Versus Mefloquine for the Treatment of Uncomplicated Malaria in Africa
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0661134
Record Dates: First submitted 2004-05-12; First posted 2004-05-14 (Estimated); Last update posted 2011-05-11 (Estimated); Status verified 2011-05

CONDITIONS: Malaria, Falciparum
MeSH Terms: conditions — Malaria, Falciparum | interventions — Azithromycin; Chloroquine; Mefloquine

INTERVENTIONS:
Drug: Azithromycin/Chloroquine
Drug: Mefloquine

SUMMARY:
The primary objective is to confirm the hypothesis that azithromycin plus chloroquine is non-inferior to mefloquine for the treatment of symptomatic, uncomplicated malaria due to P. falciparum.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent of the subject or a legally authorized representative
* Females and males
* >= 18 years of age with uncomplicated, symptomatic malaria as indicated by the presence of both of the following: a.) Blood smears positive for Plasmodium falciparum monoinfection, with asexual parasitemia between 1000 -100,000 parasites/mL b.) Fever or history of fever (>= 38.5 C/101.2 F rectal or tympanic; >= 37.5 C/99.5 F axillary or >= 38 C/100.4 F oral) within the prior 24 hours
* Serum glucose >= 60 mg/dL (by fingerstick or peripheral blood collection)
* Rapid diagnostic test (Binax NOW ICT) positive for P. falciparum
* Subjects must be willing to be treated in the inpatient setting for a minimum of three days
* Women of childbearing potential must have a negative urine gonadotropin prior to entry into the study and must agree to use adequate contraception during the entire study

Exclusion Criteria:

* Severe or complicated malaria including subjects with any of the following: a.) Impaired consciousness (e.g. obtundation, unarousable coma), seizures (any seizure within 24 hours prior to enrollment) or abnormal neurologic exam suggestive of severe or complicated malaria b.) Hemoglobinuria c.) Jaundice d.) Respiratory distress (respiratory rate >= 30/min) e.) Persistent vomiting f.) Hematuria, as reported by the patient
* Presence of non-falciparum species on microscopy
* Pregnant or breast-feeding women
* History of allergy to or hypersensitivity to azithromycin or any macrolide, mefloquine or related compounds (e.g. quinine and quinidine), or chloroquine
* Known or suspected folate deficiency
* Known history of blood dyscrasias (e.g., megaloblastic anemia, agranulocytosis, aplastic anemia, thrombocytopenia, leukopenia, neutropenia, hemolytic anemia)
* Known G-6PD deficiency
* History of epilepsy or psoriasis
* History of treatment with any antimalarial drug (chloroquine, quinine, mefloquine, Malarone, SP, artemisinin compounds) or antibacterial with known antimalarial activity (macrolides, doxycycline, clindamycin) within 2 weeks prior to enrollment into the study
* Known or suspected cardiovascular, hepatic or renal abnormality that in the opinion of the Investigator would place the subject at increased risk to participate in the study. The following findings are specific exclusions: a.) Serum creatinine >2.0 x ULN b.) ALT and/or AST >3 x ULN
* Active depression or a recent history of depression, generalized anxiety disorder, psychosis, schizophrenia or other major psychiatric disorders
* Inability to swallow oral medication in tablet form
* Treatment with other investigational drugs within 30 days prior to enrollment into the study
* Alcohol and/or any other drug abuse
* Requirement to use medication during the study that might interfere with the evaluation of the study drug
* Specific systemic diseases or other medical conditions that would interfere with the evaluation of the therapeutic response or safety of the study drug
* Inability to comprehend and/or unwillingness to follow the study protocol
* Prior participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2004-06; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Parasite clearance

SECONDARY OUTCOMES:
tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- Pfizer Investigational Site, Navrongo, Ghana
- Pfizer Investigational Site, Bamako, Mali
- Uganda (2):
  - Pfizer Investigational Site, Jinja
  - Pfizer Investigational Site, Kampala
- Pfizer Investigational Site, Ndola, Zambia
- Pfizer Investigational Site

REFERENCES:
- [Derived] Sagara I, Oduro AR, Mulenga M, Dieng Y, Ogutu B, Tiono AB, Mugyenyi P, Sie A, Wasunna M, Kain KC, Djimde AA, Sarkar S, Chandra R, Robbins J, Dunne MW. Efficacy and safety of a combination of azithromycin and chloroquine for the treatment of uncomplicated Plasmodium falciparum malaria in two multi-country randomised clinical trials in African adults. Malar J. 2014 Nov 25;13:458. doi: 10.1186/1475-2875-13-458. PMID 25425434
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661134&StudyName=Azithromycin+Plus+Chloroquine+Versus+Mefloquine+for+the+Treatment+of+Uncomplicated+Malaria+in+Africa